CLINICAL TRIAL: NCT00680563
Title: An Open Label Study of the Safety, Tolerability and Effect on Hemoglobin Levels of Once-monthly Subcutaneous Mircera in Predialysis Patients With Chronic Renal Anemia Not Currently Treated With ESA.
Brief Title: A Study of Once-Monthly Subcutaneous Mircera for the Treatment of Chronic Renal Anemia in Pre-Dialysis Patients Not Currently Treated With ESA.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21467
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — sc every month (starting dose 1.2 micrograms/kg)

SUMMARY:
This single arm study will assess the efficacy and safety of subcutaneous Mircera for the correction and maintenance of hemoglobin levels in predialysis patients with renal anemia who are not currently treated with ESA. Eligible patients will receive monthly subcutaneous injections at an initial recommended dose of 1.2 micrograms/kg. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* no ESA therapy during previous 3 months;
* adequate iron status;
* rapid chronic kidney disease progression.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension requiring hospitalization in previous 6 months;
* significant acute or chronic bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Mean change in Hb concentration between baseline and Efficacy Evaluation Period (EEP). | Week 32

SECONDARY OUTCOMES:
Time to achievement of response | Throughout study
Percentage of patients whose Hb concentration remains within range 10.0-12.0g/dL | Throughout study
Percentage of patients whose average Hb concentration is within range 10.0 - 12.0g/dL | Throughout study
Mean time spent in Hb range of 10.0 - 12.0g/dL | Throughout study
Percentage of patients requiring dose adjustments; incidence of RBC transfusions; time to initiation of renal replacement therapy. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Argentina (3):
  - Buenos Aires
  - La Plata
  - San Miguel de Tucumán
- Brazil (5):
  - Blumenau
  - Botucatu
  - Curitiba
  - Rio de Janeiro
  - São Paulo
- Santiago, Chile
- Colombia (4):
  - Barranquilla
  - Cali
  - Envigado
  - Medellín
- San José, Costa Rica
- Quito, Ecuador
- Guatemala City, Guatemala
- Panama City, Panama
- Peru (2):
  - Lima
  - San Isidro
- Caracas, Venezuela